CLINICAL TRIAL: NCT04370496
Title: Safety Of Laparoscopic or Robotic Radical Hysterectomy Using Endoscopic sTapler for Inhibiting tumOr Spillage of Cervical Neoplasms (SOLUTION): a Phase II Study
Brief Title: Safety of Minimally Invasive Surgery Using Endoscopic Stapler in Early Stage Cervical Cancer Patients (SOLUTION)
Acronym: SOLUTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB No. 2002-101-1103
Record Dates: First submitted 2020-04-19; First posted 2020-05-01 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Cervical Cancer Stage IB1; Minimally Invasive Surgery
Keywords: Cervical cancer; Cervical Cancer Stage IB1; Minimally invasive surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will undergo surgery for early stage cervical cancer. They will receive either laparoscopic or robotic radical hysterectomy using an endoscopic stapler. The efficacy and safety of this surgical technique will be compared to that of open radical hysterectomy studied in previous trials.
Masking Description: All patients enrolled in this clinical trial will undergo radical hysterectomy through minimally invasive surgery using an endoscopic stapler which both cuts and simultaneously sutures the open vaginal stump.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOLUTION group (Experimental): Patients enrolled in this clinical trial will undergo radical hysterectomy through minimally invasive surgery using an endoscopic stapler which both cuts and simultaneously sutures the open vaginal stump.
  Interventions: Procedure: Minimally invasive surgery using endoscopic stapler

INTERVENTIONS:
Procedure: Minimally invasive surgery using endoscopic stapler — Radical hysterectomy by minimally invasive surgery (laparoscopic or robotic) will be done with the help of an endoscopic stapler in cutting and suturing the uterine cervix.

SUMMARY:
The SOLUTION trial aims to show the efficacy and safety of performing radical hysterectomy by minimally invasive surgery using an endoscopic stapler in patients with cervical cancer stage IB1 (FIGO staging 2009) and thus to prove that minimally invasive surgery is non-inferior to open surgery.

DETAILED DESCRIPTION:
Cervical cancer is the 4th most common gynecologic cancer and treatment in early stages consists of surgery, chemotherapy, or radiation therapy. Surgical methods are simple or radical hysterectomy and pelvic and para-aortic lymph node dissection either done in an open manner or minimally invasive surgery (robotic or laparoscopic). However, a phase III cinical trial in 2018 comparing the safety and efficacy between minimally invasive surgery and open surgery in performing radical hysterectomy, 'Laparoscopic Approach to Cervical Cancer' (LACC), showed that open surgery is safer than minimally invasive surgery. Possible causes of such results are as follows:

1. Carbon dioxide is supplied during laparoscopic operations to maintain capnoperitoneum, which can cause the implantation and proliferation of tumor cells exposed to the peritoneal cavity.
2. Insertions of uterine manipulators into the endometrial cavity is commonly done, which can cause tumor cells to travel to both salpinges.
3. Tumor cells can be exposed to the peritoneal cavity when the cervix is exposed during intracorporeal colpotomy.
4. Tumor cells exposed to the peritoneal cavity can travel upwards when the patient's position is maintained in the Trendelenburg position during minimally invasive operations, leading to distant metastasis.

Based on the above-mentioned hypothesis, the following methods could be applied to minimize the exposure of tumor cells to the peritoneal cavity.

1. The application of a vaginal tube instead of a uterine manipulator to prevent tumor cells from traveling to the salpinges.
2. The ligation of both salpinges prior to insertion of a vaginal tube to block the travel of tumor cells.
3. The performance of extracorporeal colpotomy instead to prevent the exposure of tumor cells inside the peritoneal cavity.

Although it would be favorable to perform all the forementioned methods, extracorporeal colpotomy is difficult to perform especially in menopausal patients with atrophic vaginitis or patients with no sexual experience. Thus, an alternative method is to use an endoscopic stapler which can simultaneously cut and suture the cervix into a vaginal stump, which can prevent tumor cells from being exposed to the peritoneal cavity.

In conclusion, this clinical trial aims to show the efficacy and safety of performing radical hysterectomy by minimally invasive surgery using an endoscopic stapler in patients with cervical cancer stage IB1 (FIGO staging 2009) and thus to prove that minimally invasive surgery is non-inferior to open surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 20 years or older
* Histologically confirmed primary squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the uterine cervix
* Patients with FIGO stage IB1 (FIGO staging 2009)

  : stromal invasion>5 mm or 7 mm <lesion size ≤4 cm
* Patients undergoing either type B or C hysterectomy (Querleu-Morrow classification)
* Patients with normal bone marrow, renal and hepatic function

  * WBC > 3.0x10^9 cells/L
  * Platelets > 100x10^9 cells/L
  * Serum creatinine ≤1.5 mg/dL
  * Serum total bilirubin <1.5 x normal range and AST/SGOT or ALT/SGPT <3 x normal range
* ECOG performance status 0 or 1
* Synchronous cancer with no evidence of recurrence during the past 5 years
* Informed consent of patient

Exclusion Criteria:

* Any histological type other than squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the uterine cervix
* Tumor size greater than 4 cm
* Patients with FIGO less than stage IA2 or greater than IB2 (FIGO staging 2009)

  * stromal invasion ≤5 mm and lesion size ≤7 mm (less than IA2)
  * or lesion size> 4 cm (greater than IB2)
* Patients with evidence of metastatic disease by conventional imaging studies, enlarged pelvic or aortic lymph nodes greater than 2 cm, or histologically positive lymph nodes
* Patients in pregnancy
* Patients with a history of pelvic or abdominal radiotherapy
* Patients with contraindication of surgery (serious concomitant systemic disorders incompatible with the study to be decided at the discretion of the investigator)
* Patients who agree to intra-operative lymphatic mapping (IOLM) must not have:

  * Known allergies to triphenylmethane compounds
  * History of retroperitoneal surgery.
  * History of pelvic irradiation.
  * Cold knife or LEEP cone biopsy within 4 weeks of enrollment

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible patients must be diagnosed with cervical cancer, limiting eligibility to only females.
Enrollment: 124 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
4.5 year disease-free survival [DFS] rate | Examined at post-operative 4.5 years
  Probability of no recurrence from the day of surgery until post-operative 4.5 years

SECONDARY OUTCOMES:
4.5 year overall survival [OS] rate | Examined at post-operative 4.5 years
  Rate of survival from the day of surgery until post-operative 4.5 years
Pattern of recurrence sites | Examined every 3 months during post-operative 1 year, every 2 months during post-operative 2 years, and every 6 months during post-operative 4.5 years
  Anatomical site of recurrent cancer according to imaging modalities
Morbidity | Examined during operation and post-operative 4 and 6 weeks.
  Intra-operative and post-operative complications occurring in less than post-operative 4 weeks and between post-operative 4 and 6 weeks. Other morbidity include estimated blood loss during surgery, post-operative pain and amount of analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, M.D. Ph.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Division of Gynecologic Oncology, Department of Obstetrics and Gynecology, Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: Undecided
The plan whether to share IPD will be decided once enrollment of the clinical trial starts.

REFERENCES:
- [Background] Cohen PA, Jhingran A, Oaknin A, Denny L. Cervical cancer. Lancet. 2019 Jan 12;393(10167):169-182. doi: 10.1016/S0140-6736(18)32470-X. PMID 30638582
- [Background] Wood DE. National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Lung Cancer Screening. Thorac Surg Clin. 2015 May;25(2):185-97. doi: 10.1016/j.thorsurg.2014.12.003. Epub 2015 Jan 28. PMID 25901562
- [Result] Nam JH, Park JY, Kim DY, Kim JH, Kim YM, Kim YT. Laparoscopic versus open radical hysterectomy in early-stage cervical cancer: long-term survival outcomes in a matched cohort study. Ann Oncol. 2012 Apr;23(4):903-11. doi: 10.1093/annonc/mdr360. Epub 2011 Aug 12. PMID 21841155
- [Result] Park JY, Kim DY, Kim JH, Kim YM, Kim YT, Nam JH. Laparoscopic versus open radical hysterectomy in patients with stage IB2 and IIA2 cervical cancer. J Surg Oncol. 2013 Jul;108(1):63-9. doi: 10.1002/jso.23347. Epub 2013 Jun 5. PMID 23737035
- [Result] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Result] Kohler C, Hertel H, Herrmann J, Marnitz S, Mallmann P, Favero G, Plaikner A, Martus P, Gajda M, Schneider A. Laparoscopic radical hysterectomy with transvaginal closure of vaginal cuff - a multicenter analysis. Int J Gynecol Cancer. 2019 Jun;29(5):845-850. doi: 10.1136/ijgc-2019-000388. PMID 31155516
- [Result] Kim SI, Cho JH, Seol A, Kim YI, Lee M, Kim HS, Chung HH, Kim JW, Park NH, Song YS. Comparison of survival outcomes between minimally invasive surgery and conventional open surgery for radical hysterectomy as primary treatment in patients with stage IB1-IIA2 cervical cancer. Gynecol Oncol. 2019 Apr;153(1):3-12. doi: 10.1016/j.ygyno.2019.01.008. Epub 2019 Jan 12. PMID 30642625
- [Derived] Park SJ, Kong TW, Kim T, Lee M, Choi CH, Shim SH, Yim GW, Lee S, Lee EJ, Lim MC, Chang SJ, Lee SJ, Lee SH, Song T, Lee YY, Kim HS, Nam EJ. Safety and efficacy study of laparoscopic or robotic radical surgery using an endoscopic stapler for inhibiting tumour spillage of cervical malignant neoplasms evaluating survival (SOLUTION): a multi-centre, open-label, single-arm, phase II trial protocol. BMC Cancer. 2022 Mar 26;22(1):331. doi: 10.1186/s12885-022-09429-z. PMID 35346103
- [Derived] Mun J, Park SJ, Yim GW, Chang SJ, Kim H; Trial Monitoring Committee of SOLUTION trial. Solution to prevent tumor spillage in minimally invasive radical hysterectomy using the endoscopic stapler for treating early-stage cervical cancer: Surgical technique with video. J Gynecol Obstet Hum Reprod. 2021 Dec;50(10):102211. doi: 10.1016/j.jogoh.2021.102211. Epub 2021 Sep 1. PMID 34481135